CLINICAL TRIAL: NCT02821936
Title: Study of the Interest of the Parametric Imaging in Positron Emission Tomography on the Recurrence Prognosis at One Year in Patient With Non Small Cell Lung Cancer
Brief Title: Parametric Imaging in Positron Emission Tomography for Patient With Lung Cancer
Acronym: PARAPET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB15.03
Record Dates: First submitted 2016-06-20; First posted 2016-07-04 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: positron emission tomography; parametric imaging; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parametric Imaging (Experimental): one parametric PET at the inclusion and one at 42 Gray after the beginning of radiotherapy.
  Two PET scans at 3 months and one year after inclusion
  Interventions: Procedure: Parametric Imaging

INTERVENTIONS:
Procedure: Parametric Imaging — 2 parametric PET (one at the inclusion and one at 42 gray of the beginning of radiotherapy)

SUMMARY:
The purpose of this study is to evaluate the concordance between Positron E mission tomography parametric imaging versus standard PET for the 1 year prognosis of patients with NSCLC treated by radiochemotherapy.

The ancillary study will evaluate the interest of parametric PET imaging during the treatment (around 42 Gray) to detect the local relapse of the lesion in order to propose a treatment re-planification or intensification (not realized on the present study).

DETAILED DESCRIPTION:
In oncology, Positron Emission Tomography imaging with 18Fluor-FDG quantifies glucose metabolism lesions. Conventionally, the metabolism is quantified using the Standard Uptake Value (SUV) from a static acquisition obtained 60 minutes post-injection. Some teams reported SUV variation coefficients as high as 30% in NSCLC lesions for repeated PET examinations in patients without treatment. Moreover, information regarding the binding kinetics of 18Fluor-FDG by tumor cells is not accessible through this method.

Much more elaborated FDG quantification methods and considered as reference methods exist in PET imaging (compartmental analysis, Patlak). Simplified kinetic methods have also been proposed which correlate better with Patlak reference method than the conventional SUV. The investigators proposed a new methodological approach to obtain the parametric information in PET. This approach allows to define new indexes (average percentage of FDG-metabolized or not metabolized; time required to metabolize 80% of FDG). The approach has been clinically evaluated in a pilot study for the differentiation between benign and paraganglioma lesions.

Tsuchida observed that the parametric PET imaging allowed histological differentiation of subtypes of lung tumors, reflecting the difference in glucose transporters and hexokinase between adenocarcinoma and squamous cell carcinoma. Xue et al showed that the FDG uptake (based on the only SUV) could be a tool to predict the subtype and thus tumor staging in patients suffering from NSCLC.

The investigators can then hypothesize that some subtype of lung tumor, with increased proliferation rate (kinetic indexes k3, Ki or other parameters offered by our previous work), will be more sensitive to radiotherapy and thus the evaluation of tumor subtype by PET would allows radiotherapy adaption accordingly.

This study is a preliminary methodological study , strictly descriptive and will only assess the comparison of measurements obtained on a parametric imaging and imaging "static" in patients suffering from NSCLC . The measures of the uptake and volumes estimated by two approaches will be correlated and compared with the 1 year clinical outcome (primary objective).

An ancillary study will assess the relevance of the approach to detect, at the tumor level , an early recurrence of the disease. For this, the images acquired during the radiotherapy treatment (at 42Gy) will be analyzed retrospectively and the correlation with the images to 3 months or 1 year of relapsing patients will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient
* Age over 18 years old
* Histological evidence of non-small cell lung cancer
* Treatment by curative intent radio-chemotherapy based on platinum salt
* Stage superior or equal to T2a
* Tumour FDG uptake higher than mediastinal background noise on FDG PET/CT
* Affiliated or beneficiary of a social benefit system

Exclusion Criteria:

* Histology other than non-small cell lung cancer
* Patient without measurable target
* Absence of FDG uptake on FDG-PET/CT scan
* Previous neoplastic disease of less than 2 years duration or progressive
* Pregnant women or women of child-bearing potential or breast feeding mothers
* World Health Organisation scale superior or equal to 2
* Adult subjects who are under protective custody or guardianship
* Patient unable to comply with the specific obligations of the study (geographic, social or physical reasons) Uncontrolled diabetes with blood glucose ≥10 mmol/L, Hypersensitivity to the active substance (FDG) or to any of the excipients, Patients unable to understand the purpose of the study (language, etc.)
* Unaffiliated or not beneficiary of a social benefit system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07-13 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Prognosis of recurrence | one year
  Comparison between parametric Imaging and standard Imaging in PET for the diagnosis of recurrence

SECONDARY OUTCOMES:
analysis method of Parametric Imaging quantification determination | one year
  Determinate a method of analysis of the quantification of the parametric imaging
recurrence-free survival predictive value determination | 3 months
  Evaluate the predictive value of the technique of parametric Imaging on the recurrence-free survival at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Vera, MD, Principal Investigator — Centre Henri Becquerel
Locations (2):
- France (2):
  - APHM, Marseille
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colard E, Delcourt S, Padovani L, Thureau S, Dumouchel A, Gouel P, Lequesne J, Ara BF, Vera P, Taieb D, Gardin I, Barbolosi D, Hapdey S. A new methodology to derive 3D kinetic parametric FDG PET images based on a mathematical approach integrating an error model of measurement. EJNMMI Res. 2018 Nov 15;8(1):99. doi: 10.1186/s13550-018-0454-9. PMID 30443801